CLINICAL TRIAL: NCT00126594
Title: A Phase II Clinical Trial to Evaluate the Efficacy of BAY 43-9006 With or Without Low Dose Interferon in Metastatic Renal Cell Carcinoma
Brief Title: Sorafenib Tosylate With or Without Recombinant Interferon Alfa-2b in Treating Patients With Metastatic Kidney Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02910; NCI-2012-02910 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000437796; 2004-0526 (Other: M D Anderson Cancer Center); 6629 (Other: CTEP); N01CM62202 (NIH); P30CA016672 (NIH)
Record Dates: First submitted 2005-08-02; First posted 2005-08-04 (Estimated); Results first posted 2016-09-16 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-07

CONDITIONS: Clear Cell Renal Cell Carcinoma; Recurrent Renal Cell Carcinoma; Stage IV Renal Cell Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Sorafenib; Introns; Interferon alpha-2

ARMS (2):
- Sorafenib Tosylate (Experimental): Arm I: Oral Sorafenib 400 mg twice daily on days 1-28.
  Interventions: Drug: Sorafenib Tosylate; Other: Laboratory Biomarker Analysis
- Sorafenib Tosylate, Recombinant interferon alfa-2b (Experimental): Arm II: Sorafenib as in Arm I and low-dose Interferon alfa-2b 0.5 million units subcutaneously twice daily on days 1-28.
  Interventions: Drug: Sorafenib Tosylate; Biological: Recombinant Interferon Alfa-2b; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Sorafenib Tosylate — Given orally 400 mg orally (PO) every 12 hours
  Other Names: BAY 54-9085; Nexavar; SFN; BAY 43-9006
Biological: Recombinant Interferon Alfa-2b — Given subcutaneously (SC) 0.5 million with +/- 5 % variance (0.475 MU - 0.525 MU); Dose level 0: 0.5 X 10^6 international units twice daily
  Other Names: Alfatronol; Glucoferon; Heberon Alfa; Sch 30500; Urifron; IFN
  Arms: Sorafenib Tosylate, Recombinant interferon alfa-2b
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This randomized phase II trial is studying sorafenib and interferon alfa-2b to see how well they work compared to sorafenib alone in treating patients with metastatic kidney cancer. Sorafenib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Interferon alfa-2b may interfere with the growth of tumor cells. Sorafenib and interferon alfa-2b may also block blood flow to the tumor. Giving sorafenib together with interferon alfa-2b may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Efficacy of Bay 43-9006 with or without low dose interferon by evaluating response rate in MRCC.

II. Toxicities of Bay 43-9006 with or without low dose interferon in MRCC.

SECONDARY OBJECTIVES:

I. Progression free survival. II. Duration of response. III. Overall Survival.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

Arm I: Patients receive oral sorafenib twice daily on days 1-28.

Arm II: Patients receive sorafenib as in arm I and low-dose interferon alfa-2b subcutaneously twice daily on days 1-28.

In both arms, courses repeat every 28 days in the absence of progressive disease or unacceptable toxicity.

Tissue samples are analyzed for single nucleotide polymorphisms (SNP) patterns via genotyping.

After completion of study treatment, patients are followed every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically confirmed metastatic clear cell RCC
* Patients must have measurable disease, defined as a lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) and measures >= 20 mm with conventional techniques or >= 10 mm with spiral CT scan
* ECOG performance status =< 1
* Absolute neutrophil count >= 1,500/μL
* Platelets >= 100,000/μL
* Hgb > 9.0 g/dL (may be transfused or receive epoetin alfa [e.g., Epogen®] to maintain or exceed this level)
* Total bilirubin =< 2.0 mg/dl
* Albumin > 3.0 g/dL
* Serum creatinine =< 2.0 mg/dl
* AST(SGOT) and/or ALT (SGPT) =< 2.5 X institutional upper limit of normal for subjects without evidence of liver metastases
* AST(SGOT) and/or ALT (SGPT) =< 5 X institutional upper limit of normal for subjects with documented liver metastases
* Female patients of childbearing potential must have a normal plasma beta human chorionic gonadotropin (βHCG) within 24 hours prior to enrolling in the study due to the possible teratogenic effect; however, patients will be eligible if their βHCG elevation is consistent with malignancy rather than pregnancy
* Patients of child fathering or childbearing potential must agree to practice a form of medically acceptable birth control while on study
* Patients must give written informed consent prior to initiation of therapy, in keeping with the policies of the institution; patients with a history of major psychiatric illness must be judged able to fully understand the investigational nature of the study and the risks associated with the therapy; the only approved consent is attached to this protocol
* Patients must have ability to comply with study and/or follow-up procedures
* Patients must be able to swallow pills

Exclusion Criteria:

* No prior malignancy is allowed, except for non-melanoma skin cancer, in situ carcinoma of any site, or other cancers for which the patient has been adequately treated and disease free for 5 years
* Patients must not have received any systemic anticancer therapy for renal cell carcinoma; patients must not have received any radiotherapy for renal cell carcinoma within 4 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients must not be scheduled to receive another experimental drug while on this study; patients are permitted to be on concomitant bisphosphonates
* Patients must not have a primary brain tumor, any brain metastases, leptomeningeal disease, seizure disorders not controlled with standard medical therapy, or history of stroke
* Patients must not have active acute infections that could be worsened by anticancer therapy or interfere with this study
* Patients must not have clinically significant cardiovascular disease, myocardial infarction within the past year (unstable angina), New York Heart Association (NYHA) Grade II or greater congestive heart failure, serious cardiac dysrhythmia refractory to medical management, or peripheral vascular disease (Grade II or greater)
* Patients must not have uncontrolled hypertension
* Patients must not have history of other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that might affect the interpretation of the results of the study or render the subject at high risk from treatment complications
* Pregnant women are excluded from this study because BAY 43-9006 is a kinase inhibitor agent with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with BAY 43-9006, breastfeeding should be discontinued if the mother is treated with BAY 43-9006
* Patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy; therefore, HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with BAY 43-9006; appropriate studies will be undertaken in patients receiving combination anti-retroviral therapy when indicated
* Patients must not have a clinical history of coagulopathy, bleeding diathesis or thrombosis; patients must not be on therapeutic anticoagulation; prophylactic anticoagulation (ie low dose warfarin) of venous access devices is allowed provided that INR >= 1.5 is due to warfarin therapy; other patients with an INR >= 1.5 are excluded
* Patients must not have a history of severe depression
* Concomitant treatment with rifampin, St. John's wort, and the cytochrome p450 enzyme-inducin antiepileptic drugs (phenytoin, carbamazepine or Phenobarbital)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2005-06; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Jonasch, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Aldin A, Besiroglu B, Adams A, Monsef I, Piechotta V, Tomlinson E, Hornbach C, Dressen N, Goldkuhle M, Maisch P, Dahm P, Heidenreich A, Skoetz N. First-line therapy for adults with advanced renal cell carcinoma: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 May 4;5(5):CD013798. doi: 10.1002/14651858.CD013798.pub2. PMID 37146227
- [Derived] Gatto F, Bratulic S, Jonasch E, Limeta A, Maccari F, Galeotti F, Volpi N, Lundstam S, Nielsen J, Stierner U. Plasma and Urine Free Glycosaminoglycans as Monitoring and Predictive Biomarkers in Metastatic Renal Cell Carcinoma: A Prospective Cohort Study. JCO Precis Oncol. 2023 Feb;7:e2200361. doi: 10.1200/PO.22.00361. PMID 36848607
- [Derived] Ho TH, Liu XD, Huang Y, Warneke CL, Johnson MM, Hoang A, Tamboli P, Wang F, Jonasch E. The impact of FGFR1 and FRS2alpha expression on sorafenib treatment in metastatic renal cell carcinoma. BMC Cancer. 2015 Apr 18;15:304. doi: 10.1186/s12885-015-1302-1. PMID 25900027

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: June 23, 2005 to June 28, 2007. All recruitment done at The University of Texas (UT) MD Anderson Cancer Center.
Period: Overall Study
Arm/Group | Sorafenib Tosylate | Sorafenib Tosylate, Recombinant Interferon Alfa-2b
Started | 40 | 40
Completed | 1 | 3
Not Completed | 39 | 37
Not completed — Ineligible | 2 | 0
Not completed — Withdrawal by Subject | 0 | 4
Not completed — Physician Decision | 1 | 3
Not completed — Adverse Event | 7 | 5
Not completed — Non-compliance | 0 | 1
Not completed — Disease Progression | 29 | 24

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sorafenib Tosylate | Sorafenib Tosylate, Recombinant Interferon Alfa-2b | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Full Range); unit: years] | 62.4 [45 to 83] | 60.7 [43 to 81] | 62.0 [43 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 11 | 19
  Male | 32 | 29 | 61
Region of Enrollment [Number; unit: participants]
  United States | 40 | 40 | 80
ECOG (Performance Status) [Number; unit: participants] — Eastern Cooperative Oncology Group (ECOG) Scale used to assess how a participant's disease is progressing, assess how the disease affects the daily living abilities of the participant, and determine appropriate treatment and prognosis. Scale runs from 0 to 5, with 0 denoting perfect health and 5 death.
  participants
    0 | 25 | 25 | 50
    1 | 15 | 15 | 30
Nephrectomy [Number; unit: participants] — Number of participants who had nephrectomy
  participants
    Yes | 40 | 39 | 79
    No | 0 | 1 | 1
Memorial Sloan-Kettering Cancer Center (MSKCC) Prognostic Risk [Number; unit: participants] — MSKCC risk system stratifies participants poor, intermediate and favorable-risk categories based on number of adverse clinical/laboratory parameters present. Poor prognostic factors include Karnofsky performance status <80, time from diagnosis to treatment <12 months, serum lactate dehydrogenase >1.5-times upper limit of normal, corrected serum calcium >10.0 mg/dl & hemoglobin <lower limit of normal. Favorable-risk group have no poor prognostic factors, intermediate-risk category have 1 or 2 adverse prognostic factors, & participants with poor-risk have >2 poor prognostic factors.
  participants
    Low | 21 | 20 | 41
    Intermediate | 19 | 18 | 37
    Poor | 0 | 2 | 2
Number of Metastatic Sites [Number; unit: participants]
  One | 13 | 14 | 27
  Two | 17 | 20 | 37
  Three or More | 10 | 6 | 16
Sites of Metastatic Disease [Number; unit: participants] — Number of participants with metastatic tumor sites in the noted locations for each study arm population.
  participants
    Lung | 33 | 30 | 63
    Lymph Nodes | 20 | 15 | 35
    Liver | 3 | 5 | 8
    Bone | 5 | 6 | 11
    Other | 19 | 19 | 38

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) Evaluated Using Response Evaluation Criteria in Solid Tumors (RECIST)
Description: ORR defined as participants with Complete Response (CR) and Partial Response (PR) as defined by RECIST criteria: Complete Response (CR): Disappearance all target lesions. Partial Response (PR): >30% decrease in sum of longest diameter (LD) of target lesions, reference baseline sum LD. Progressive Disease (PD): >20% increase in sum of LD of target lesions, reference smallest sum LD recorded since treatment started or appearance of one or more new lesions. Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, reference smallest sum LD since treatment started. Radiologic testing for progressive disease repeated every 8 weeks.
Time Frame: Tumor restaging performed at 8 weeks following baseline, responding or stable participants restaged at 8 week intervals, up to 12 months.
Population: Analysis performed for the intent-to-treat population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sorafenib Tosylate | Sorafenib Tosylate, Recombinant Interferon Alfa-2b
Number analyzed (Participants) | 40 | 40
percentage of participants | 30 [16.56 to 46.53] | 25 [12.69 to 41.20]

2. Secondary Outcome: Selected Grade 3-4 Adverse Events Using NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0
Description: Adverse events graded using the CTCAE version 4.0 tabulated by treatment arm within either toxicity grade for the treatment period. Treatment-related toxicity (acute and cumulative) performed every 8 weeks during the first year.
Time Frame: Up to 12 months of treatment
Population: All participants were included in adverse event reporting per intent to treat analysis.
Measure: Number; unit: participants
Arm/Group | Sorafenib Tosylate | Sorafenib Tosylate, Recombinant Interferon Alfa-2b
Number analyzed (Participants) | 40 | 40
participants
  Fatigue | 10 | 13
  Diarrhea | 13 | 8
  Hand-Foot Syndrome | 10 | 7
  Hyperuricemia | 12 | 3
  Hyperamylasemia or Lipasemia | 5 | 4
  Dyspnea | 4 | 4
  Hypophosphatemia | 3 | 5
  Neutropenia | 0 | 6
  Hypertension | 2 | 3
  Nausea and vomiting | 1 | 3
  Rash/Desquamation | 2 | 2
  Proteinuria | 1 | 2
  Syncope (Fainting) | 0 | 3
  Weight Loss | 0 | 3
  Transaminitis | 0 | 3
  Hyponatremia | 2 | 1
  Nonneutropenic Infection | 2 | 0
  Sensory Neuropathy | 1 | 1
  Cardiac Ischemia/Infarction | 1 | 0
  Appendicitis | 1 | 0
  Pancreatitis | 1 | 0
  Adrenal Insufficiency | 0 | 1
  Reversible Posterior Leukonencephalopathy | 0 | 1
  Small Bowel Obstruction | 1 | 0
  Pneumonitis | 1 | 0

3. Secondary Outcome: Progression-free Survival
Description: Progression free survival (PFS) is defined as the time interval from the start of protocol therapy to death or disease progression.
Time Frame: From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
Population: All participants were included per intent to treat analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sorafenib Tosylate | Sorafenib Tosylate, Recombinant Interferon Alfa-2b
Number analyzed (Participants) | 40 | 40
Months | 7.39 [5.52 to 9.20] | 7.56 [5.19 to 11.07]

4. Secondary Outcome: Median Overall Survival (OS)
Description: Overall survival defined as the time interval from the start of protocol therapy to death or date of last follow-up if alive.
Time Frame: From the start of protocol therapy to death or date of last follow-up, up to 36 months
Population: Participants who die of unrelated cause during therapy or are lost to follow-up were censored. Median OS was not reached in Arm 1: Sorafenib as subjects experienced different events that made further follow-up impossible i.e. disease complications, death or lost to follow-up so overall survival data was not attainable.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sorafenib Tosylate | Sorafenib Tosylate, Recombinant Interferon Alfa-2b
Number analyzed (Participants) | 40 | 40
Months | NA [NA to NA] — Median OS nor limits attained due to censoring of participants who died of unrelated cause during therapy or were lost to follow-up. | 27.04 [22.31 to NA] — Upper limit not attained due to censoring of participants who died of unrelated cause during therapy or were lost to follow-up.

5. Secondary Outcome: Duration of Response for Participants With Stable Disease (N=37) Following Treatment
Description: Duration of response for participants with disease stabilization following treatment as measured from the date response is confirmed to the date of disease progression, first assessed up to 8 weeks (2 cycles) following start of treatment. The duration of a Stable Disease (SD) response is measured from the time measurement criteria are met for that specific SD response until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started). Repeat radiologic studies (CT, MRI, Chest x-ray and bone scan as indicated) to evaluate disease progression or response every 8 weeks.
Time Frame: From the date response is confirmed to the date of disease progression, up to 12 months
Population: Combined analysis reflects overall stable disease duration e.g. duration of benefit for stable disease cases without being affected by the median duration not attainable for the separate arms; 37 participants in the two arms met "Stable Disease" criteria: 17 in Sorafenib alone (Arm I) and 20 in the Sorafenib Plus Interferon group (Arm II).
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Sorafenib Tosylate or Sorafenib Plus Interferon: Arm I: Oral Sorafenib 400 mg twice daily on days 1-28 and Arm II: Sorafenib as in Arm I and low-dose Interferon alfa-2b 0.5 million units subcutaneously twice daily on days 1-28.
Arm/Group | Sorafenib Tosylate or Sorafenib Plus Interferon
Number analyzed (Participants) | 37
Months | 5.7 [3.7 to 8.4]

6. Post Hoc Outcome: Best Overall Response for Participants
Description: Best overall response is the best response recorded from the start of the treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the treatment started). The participant's best response assignment will depend on the achievement of both measurement and confirmation criteria as defined by RECIST: Complete Response (CR): Disappearance all target lesions. Partial Response (PR): >30% decrease in sum of longest diameter (LD) of target lesions, reference baseline sum LD. Progressive Disease (PD): >20% increase in sum of LD of target lesions, reference smallest sum LD recorded since treatment started or appearance of one or more new lesions. Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, reference smallest sum LD since treatment started. Radiologic testing for progressive disease repeated every 8 weeks.
Time Frame: From the date response is confirmed to the date of disease progression, first assessed 2 months (8 weeks) following start of treatment and reassessed up to 36 months (on average reassessed 12 months or less).
Population: All participants were included per intent to treat analysis.
Measure: Number; unit: participants
Arm/Group | Sorafenib Tosylate | Sorafenib Tosylate, Recombinant Interferon Alfa-2b
Number analyzed (Participants) | 40 | 40
participants
  Complete Response (CR) | 1 | 0
  Partial Response (PR) | 11 | 10
  Stable Disease (SD) | 17 | 20
  Progressive Disease (PD) | 6 | 7
  Inevaluable | 5 | 3

ADVERSE EVENTS:
Time Frame: Adverse event reporting from time of first intervention to follow up 30 days beyond last intervention. Overall study period: June 2005 to August 2013.
Description: Revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 utilized for AE reporting until September 30, 2010. CTCAE version 4.0 utilized beginning October 1, 2010.
Arm/Group | Sorafenib Tosylate | Sorafenib Tosylate, Recombinant Interferon Alfa-2b
Serious Adverse Events (participants affected / at risk) | 29/40 | 30/40
Other Adverse Events (participants affected / at risk) | 40/40 | 40/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sorafenib Tosylate (N=40) | Sorafenib Tosylate, Recombinant Interferon Alfa-2b (N=40)
Death (General disorders) | 27 (27) | 29 (29)
Pancreatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 6 (12) | 2 (2)
Serum amylase increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Lipase Increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sorafenib Tosylate (N=40) | Sorafenib Tosylate, Recombinant Interferon Alfa-2b (N=40)
Abdominal distension (Gastrointestinal disorders) | 4 (4) | 4 (5)
Abdominal pain (Gastrointestinal disorders) | 7 (15) | 10 (12)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Metabolism and nutrition disorders) | 7 (10) | 23 (41)
Alkaline phosphatase increased (Metabolism and nutrition disorders) | 13 (19) | 11 (14)
Allergic reaction (Immune system disorders) | 0 (0) | 1 (1)
Allergic rhinitis (Immune system disorders) | 2 (3) | 3 (5)
Alopecia (Skin and subcutaneous tissue disorders) | 22 (22) | 20 (20)
Anemia (Blood and lymphatic system disorders) | 19 (30) | 30 (60)
Anorexia (Gastrointestinal disorders) | 9 (10) | 10 (17)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (21) | 7 (23)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (3) | 2 (2)
Aspartate aminotransferase increased (Metabolism and nutrition disorders) | 22 (33) | 29 (55)
Back pain (Musculoskeletal and connective tissue disorders) | 11 (20) | 13 (42)
Bladder infection (Renal and urinary disorders) | 2 (2) | 0 (0)
Bladder spasm (Renal and urinary disorders) | 1 (1) | 0 (0)
Blood bilirubin increased (Blood and lymphatic system disorders) | 9 (17) | 11 (17)
Blurred vision (Eye disorders) | 3 (3) | 5 (9)
Bone pain (Musculoskeletal and connective tissue disorders) | 6 (16) | 6 (20)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Carbon monoxide diffusing capacity decreased (Investigations) | 0 (0) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Chills (General disorders) | 0 (0) | 2 (2)
Cholesterol high (Metabolism and nutrition disorders) | 15 (25) | 7 (12)
Conduction disorder (Cardiac disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 4 (9) | 5 (11)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (18) | 11 (19)
Creatinine increased (Metabolism and nutrition disorders) | 10 (18) | 8 (15)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 3 (4) | 7 (7)
Diarrhea (Gastrointestinal disorders) | 33 (375) | 32 (382)
Dizziness (Nervous system disorders) | 2 (3) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 27 (50) | 22 (50)
Dysgeusia (Gastrointestinal disorders) | 4 (5) | 7 (7)
Dyspepsia (Gastrointestinal disorders) | 3 (4) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 16 (33) | 20 (64)
Edema limbs (General disorders) | 4 (4) | 2 (2)
Edema trunk (General disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (8) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 3 (3) | 1 (1)
Extraocular muscle paresis (Eye disorders) | 1 (1) | 0 (0)
Eye disorders (Eye disorders) | 1 (1) | 1 (4)
Eye pain (Eye disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 33 (184) | 36 (247)
Fever (Investigations) | 7 (17) | 10 (20)
Flatulence (Gastrointestinal disorders) | 7 (13) | 7 (14)
Flu like symptoms (Investigations) | 0 (0) | 3 (6)
Flushing (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Gait disturbance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal disorders (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 3 (8) | 5 (6)
Hemoglobinuria (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 3 (14)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 22 (42) | 17 (47)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 (6) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 10 (16) | 8 (12)
Hypertension (Cardiac disorders) | 16 (26) | 10 (14)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 20 (20) | 21 (49)
Hyperuricemia (Metabolism and nutrition disorders) | 24 (66) | 19 (37)
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 (5) | 6 (9)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2) | 14 (37)
Hypoglycemia (Metabolism and nutrition disorders) | 22 (42) | 3 (8)
Hypokalemia (Metabolism and nutrition disorders) | 10 (16) | 6 (9)
Hypomagnesemia (Metabolism and nutrition disorders) | 17 (37) | 21 (42)
Hyponatremia (Metabolism and nutrition disorders) | 5 (8) | 4 (7)
Hypophosphatemia (Metabolism and nutrition disorders) | 20 (36) | 20 (49)
Hypotension (Cardiac disorders) | 1 (1) | 2 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Infections and infestations - (Other) (Infections and infestations) | 5 (6) | 3 (3)
Injection site reaction (Injury, poisoning and procedural complications) | 0 (0) | 5 (8)
Insomnia (General disorders) | 0 (0) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Lipase increased (Metabolism and nutrition disorders) | 5 (9) | 5 (5)
Lung infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lymphocyte count decreased (Blood and lymphatic system disorders) | 4 (9) | 12 (51)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 14 (77) | 18 (39)
Myalgia (Musculoskeletal and connective tissue disorders) | 10 (20) | 8 (15)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 18 (57) | 24 (60)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (6) | 1 (1)
Nervous system disorders - (Other) (Nervous system disorders) | 0 (0) | 1 (1)
Neutrophil count decreased (Metabolism and nutrition disorders) | 0 (0) | 18 (47)
Non-cardiac chest pain (General disorders) | 3 (7) | 3 (4)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Otitis media (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 7 (17) | 5 (13)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 (35) | 14 (39)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 32 (77) | 31 (109)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Pancreatitis (Hepatobiliary disorders) | 0 (0) | 0 (0)
Pelvic pain (General disorders) | 0 (0) | 1 (3)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 10 (20) | 14 (42)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
Platelet count decreased (Blood and lymphatic system disorders) | 2 (2) | 21 (39)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Infections and infestations) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 16 (31) | 24 (48)
Pruritus (Skin and subcutaneous tissue disorders) | 8 (8) | 4 (6)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 30 (63) | 26 (62)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Renal and urinary disorders - (Other) (Renal and urinary disorders) | 1 (1) | 1 (2)
Reproductive system and breast disorders - (Other) (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal disorders - (Other) (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1)
Scrotal pain (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Serum amylase increased (Metabolism and nutrition disorders) | 3 (3) | 4 (4)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - (Other) (Skin and subcutaneous tissue disorders) | 11 (18) | 12 (25)
Skin infection (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Sore throat (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 1 (5) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 3 (3)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 1 (2)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (2) | 1 (1)
Tremor (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 1 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Vascular disorders - (Other) (Cardiac disorders) | 0 (0) | 2 (5)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Vomiting (Gastrointestinal disorders) | 11 (42) | 14 (34)
Watering eyes (Eye disorders) | 2 (2) | 0 (0)
Weight loss (General disorders) | 15 (27) | 21 (42)
White blood cell decreased (Metabolism and nutrition disorders) | 3 (4) | 27 (63)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less